CLINICAL TRIAL: NCT04274868
Title: Constitution of a Centralized Biological Resources Collection and Associated With a Clinical Database for Childhood Liver Tumors Diagnosed in France (Retrospective Collection From 1990 and Prospective)
Brief Title: Pediatric Hepatic Tumors
Acronym: HEPATOBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A00180-49
Record Dates: First submitted 2020-02-17; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Liver Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents with liver tumor: Patients treated after 01/01/1990 for a primary liver tumor before the age of 18.

SUMMARY:
Centralized biological collection of multicentric origin, retrospective and prospective of biological samples (tissues and fluids) taken within the framework of the diagnostic and therapeutic management of children and adolescents with liver tumor, and supported in the centers of French Society for Childhood Cancers (SFCE) with associated clinical database.

ELIGIBILITY:
Inclusion Criteria:

1. - For inclusion in the clinical database:

   * Children and adolescents (≤18 years at diagnosis) suffering from a primary liver tumor diagnosed after 01/01/1990 and treated in France
   * Informed consent to the computerization of data signed by the patient or by parents or legal representatives if he is a minor.
2. - For inclusion in the biological collection (CRB Paris Sud):

   * Additional criteria:
   * Availability of biological samples (tumor tissue, healthy tissue, plasma and / or serum).
   * Informed consent to the use of biological remains signed by the patient or by parents or legal representatives if he is a minor.
3. - For the inclusion of deceased patients:

   * Obtaining consent or failing this, seeking non-opposition to the computerization of data (for inclusion in the database) and the use of biological remains (for inclusion in the biological collection) of the patient or both parents or the legal guardian if he is a minor.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients treated after 01/01/1990 for a primary liver tumor before the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Establish a national bank of rare biological material | Up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No